CLINICAL TRIAL: NCT06831136
Title: Endoscopic Ultrasound Radiofrequency Ablation and Immunotherapy Pembrolizumab for Locally Advanced Unresectable and Metastatic Pancreatic Duct Adenocarcinoma; a Phase II Trial PANcreas CAncer RaDIofrequeNcy AbLation
Brief Title: Endoscopic Ultrasound Radiofrequency Ablation and Immunotherapy Pembrolizumab for Locally Advanced Unresectable and Metastatic Pancreatic Duct Adenocarcinoma
Acronym: PANCARDINAL-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Putao Cen, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-0437
Record Dates: First submitted 2025-01-16; First posted 2025-02-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: metastatic cancer; chemotherapy; systemic immunotherapy; pembrolizumab; neoplasms; Endoscopic Ultrasound Radiofrequency ablation (EUS-RFA)
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Neoadjuvant Therapy; Immunotherapy; pembrolizumab; Endosonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Standard of care chemotherapy + immunotherapy + EUS-RFA (Experimental)
  Interventions: Drug: Neoadjuvant Chemotherapy (NAC); Drug: Immunotherapy (pembrolizumab); Device: Endoscopic ultrasound (EUS)-guided radiofrequency ablation (RFA)

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy (NAC) — Participant will undergo 8 weeks of NAC (treating physician's choice). Possible regimens are either mFOLFIRINOX or NALIRIFOX or Gemcitabine Nab-Paclitaxel ± Cisplatin (GA+/-Cisplatin) or Capecitabine (Xeloda).
Drug: Immunotherapy (pembrolizumab) — 2-12 weeks after initial chemotherapy and after the first EUS-RFA treatment, patients will receive 400 mg every 6 weeks of pembrolizumab via infusion. Participants will be administered standard of care chemotherapy and pembrolizumab every 6 weeks.
Device: Endoscopic ultrasound (EUS)-guided radiofrequency ablation (RFA) — After 2-12 weeks of chemotherapy, patients will undergo EUS-RFA treatment 1 session every 6 weeks. Each RFA treatment will be for up to 5 cycles at 30W for 20 seconds or until there is an increase in measured impedance. After the 5th EUS-RFA, if there is clinical benefit, then patients will continue with EUS-RFA treatments until no active tumor is seen. During each session, the therapeutic gastroenterologist will evaluate if there is any tumor to undergo RFA. If no active tumor seen, then will abort RFA

SUMMARY:
The purpose of this study is to perform a pilot phase II trial to evaluate the safety and efficacy of combined EUS-RFA, chemotherapy, and systemic immunotherapy (pembrolizumab) for the treatment of locally advanced unresectable and metastatic Pancreatic ductal adenocarcinoma (mPDAC).

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to comply with the protocol for the duration of the study,including undergoing treatment and scheduled visits and examinations, including follow-up
* Biopsy-proven locally advanced unresectable or metastatic PDAC

  1. Patients who have undergone prior resection will be excluded unless there is recurrent pancreatic tumor that is amenable to EUS-RFA.
  2. If biliary metal stent is placed, during procedure of EUS-RFA, indwelling biliary metal stent will be removed during initial EUS-RFA and then replaced with plastic stent.
* Mental capacity to provide informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* At least one measurable metastatic lesion on axial imaging per Response Evaluation Criteria in Solid Tumors (RECIST) v1.
* No prior systemic therapy, including chemotherapy or chemoradiation is permitted with the following exceptions:

  1. Prior adjuvant therapy (including chemotherapy and/or radiotherapy) for pancreatic adenocarcinoma is permitted if standard of care neoadjuvant or adjuvant therapy was completed at least 3 months prior to study enrollment. Prior adjuvant therapy may include mFFX, NALIRIFOX, GA or Capecitabine (Xeloda).
  2. If started on first-line treatment for mPDAC elsewhere (i.e., not at our study site), eligible participants can have undergone 3 months of chemotherapy with stable disease before study entry. Note: Imaging done outside the site will need to be reviewed for a 2nd opinion to confirm stable disease.

  i. For patients who had prior treatment and stable disease up to 3 months and confirmed radiographically by our radiology investigators, then patients can proceed with EUS-RFA within 6-8 weeks of enrollment of study.

  c. Patients who have started chemotherapy within a 3-month timeframe are allowed.
* Absolute neutrophil count (ANC) ≥1 x 109/L
* Platelet count ≥75 x 109/L
* Albumin levels ≥3 g/dL
* Total serum bilirubin <2× upper limit of normal (ULN) unless secondary to Gilbert's Syndrome

  a. Subjects requiring biliary decompression, biliary stent, or drainage using percutaneous trans-hepatic cholangiogram are allowed (patients with a declining bilirubin status post stent placement are eligible with serum bilirubin ≤2.5 x ULN)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤3× ULN, or ≤5× ULN in cases of documented liver involvement
* Serum creatinine clearance must be ≥30 mL/minute either measured or calculated using a standard Cockcroft and Gault formula
* Prior surgery that required general anesthesia or other major surgery as defined by the Investigator must be completed at least 4 weeks before immunotherapy.

Exclusion Criteria:

* No telephone number and permanent street address
* Pregnant or breastfeeding patients; or is a male or female patient of reproductive potential who is not willing to employ effective birth control from time of screening to 90 days after the last dose
* Inmates or prisoners
* Unable to provide informed consent
* Resectable, borderline resectable PDAC.
* Known history of central nervous system (CNS) metastases
* Has a history of another primary malignancy. Patients having the following are still eligible:

  1. No active stage 4 cancer
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* Known low or absent dihydropyrimidine dehydrogenase (DPD) activity
* Use of strong inhibitors or inducers of Cytochrome P450 3A (CYP3A), CYP2C8 and UGT1A1
* History or evidence of clinically significant or uncontrolled cardiovascular, CNS,and/or other systemic disease that in the investigator's opinion would preclude participation in the study or compromise the patient's ability to give informed consent
* History of HIV or active tuberculosis (TB) (PPD response without active TB is allowed)
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of pembrolizumab hazardous (e.g., interstitial lung disease, active infections requiring antibiotics, recent hospitalization with unresolved symptoms)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Any active autoimmune disease or a documented history of autoimmune disease or history of a syndrome that required systemic steroids or immunosuppressive medications, except for vitiligo or resolved childhood asthma/atopy and the following scenarios below:

  1. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study.
  2. Physiologic doses of corticosteroids (≤10 mg/day of prednisone or its equivalent) or short pulses of corticosteroids (≤3 days) may be permitted.
  3. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  4. Patients having any chronic skin condition that does not require systemic therapy
  5. Patients without active disease in the last 5 years (allowed only after consultation with the study physician)
  6. Patients with celiac disease controlled by diet alone
* Is currently using or previously used immunosuppressive medication within 14 days before the first dose of pembrolizumab. The following medications are exceptions to this criterion:

  1. intranasal, inhaled, topical steroid, or local steroid injections (e.g., intra articular injection)
  2. Systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
  3. steroids as premedication for hypersensitivity reactions (e.g., computer tomography [CT] scan premedication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-01-20 (Estimated); Study Completion 2030-01-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy as assessed by the Overall response rate using RECIST v1.1 guidelines | From date of diagnosis to the initial date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months.
  (ORR) is defined as proportion of patients with complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From the date of the initiation of study treatment until 30 days after the last dose of study treatment, withdrawal of consent, or study termination
Incidence of serious adverse events (SAEs) | From the date of the initiation of study treatment until 30 days after the last dose of study treatment, withdrawal of consent, or study termination
Duration of response (DOR) | Every 8 weeks from the time of enrollment to the date of death due to any causes for up to 5 years
  DOR is defined as elapsed time between date of documented response (CR or PR) and date of progression or date of death from any cause.
Progression-free survival (PFS) | Every 8 weeks from the time of enrollment to the date of death due to any causes for up to 5 years
  Progression-free survival (PFS) is defined as elapsed time between start date of treatment and date of progression or date of death from any cause.
Overall survival (OS) | Every 8 weeks from the time of enrollment to the date of death due to any causes for up to 5 years
  Overall survival (OS) is defined as elapsed time between start date of treatment and date of death from any cause.
Local (distant) recurrence rate | Every 8 weeks from the time of enrollment to the date of death due to any causes for up to 5 years
  Local (distant) recurrence rate is defined as incidence rate of local (distant) recurrence
Local (distant) recurrence time | Every 8 weeks from the time of enrollment to the date of death due to any causes for up to 5 years
  Local (distant) recurrence time is defined as the elapsed time between start date of treatment and date of the first local (distant) recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Putao Cen, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No